CLINICAL TRIAL: NCT06499961
Title: The Digital Version of Holistic Healthy Life Education: A Randomized Controlled Trial
Brief Title: The Digital Version of Holistic Healthy Life Education(e2HLE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Yan Chai Hospital (Other)
Responsible Party: Principal Investigator, Dr Angela Leung, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03
Record Dates: First submitted 2024-05-07; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
Keywords: healthy lifestyle
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital version of Holistic Healthy Life Education (e2HLE) (Experimental)
  Interventions: Behavioral: Digital version of Holistic Healthy Life Education
- Waitlist-control (Other)
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: Digital version of Holistic Healthy Life Education — Participants need to attend a two-day workshop related to (1) health risk appraisal and self-care; (2) exercise, fitness and self-acupressure; (3) emotion and stress management; (4) the whole food plant-based (WFPB) diet; and (5) meditation and mindfulness practices, led by a multi-disciplinary team. Before the intervention commences, they will take pre-blood test and further receive the e2HLE with Hera Leto for three months. During the intervention, participants will attend (1) nine weekly workshops pertaining to WFPB diet, exercise, fitness and self-acupressure, and meditation and mindfulness and followed by weekly tele-counselling sessions; (2) three process evaluation practice sharing sessions in the format of focus group, making up a total of twelve sessions. The process evaluation practice sharing sessions will be audio-recorded; (3) mutual support networking platform will be held between case managers and participants within Hera Leto system.
  Arms: digital version of Holistic Healthy Life Education (e2HLE)
Other: Waitlist control — usual care first, then switch to receive the intervention
  Arms: Waitlist-control

SUMMARY:
The digital version of Holistic Healthy Life Education" (e2HLE) is a holistic, person-centric, multi-component and lifestyle modification intervention that we developed, alongside the WHO integrated care for older people (ICOPE) model and a home-based self-monitoring bio-signals system "Hera Leto". This randomized controlled trial aims to evaluate the effectiveness of e2HLE intervention for achieving weight loss and enhancing self-care and intrinsic capacity (i.e. psychological and mental wellbeing, vitality and nutritional health) as well as improving cardio-metabolic profiles (e.g. blood pressure and lipid profile) compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 years old or above,
* able to use internet and tablet;
* education level of primary or above;
* understand Chinese and speak Cantonese;
* have central obesity (waist circumference: male >90 cm, female >80 cm) and two of the following: (a) hypertension (systolic blood pressure ≥130 or diastolic blood pressure ≥85 mmHg, or treatment of previously diagnosed hypertension), (b) hyperglycemia (fasting plasma glucose ≥100 mg/dL (5.6 mmol/L) or (c) previously diagnosed type 2 diabetes), (d) hyperlipidemia (triglyceride concentrations ≥150 mg/dL (1.7 mmol/L), or treatment for this lipid abnormality); HDL cholesterol;40 mg/dL (1.03 mmol/L) in males and 50 mg/dL (1.29 mmol/L) in females, or treatment for this lipid abnormality), (e) BMI over 23; and chronic pain or bad mood caused by the psychosomatic disorder for no less than six months
* have at least 2 of the following distressing symptoms due to psychosomatic or pain and stress symptoms, including physical and mental agitation, feeling tired, often crying, feeling angry/depressed, feeling isolated from family and friends, feeling great stress, insomnia, health is worse than before.

Exclusion Criteria:

* non-Chinese nationality or can't speak Cantonese;
* participating in any cancer treatment;
* will leave Hong Kong within a short period or the next three months;
* participating in another experiment; living in or planning to live in a facility-care home;
* cognitive difficulties (SPMSQ score equal to or lower than 4);
* taking medications such as estrogenic, synthetic glucocorticoids, anti-steroids, and antiepileptic drugs which may affect cortisol levels.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-05-21 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 3 months
  Weight change from baseline to post-intervention (kg)

SECONDARY OUTCOMES:
Intrinsic capacity | 3 months
  WHO ICOPE tool including five domains: cognitive, locomotor, sensory, vision, and psychological capacity. A total score ranges from 0 to 6, a higher score indicating a poor intrinsic capacity
Heart rate variability | 3 months
  measured in milliseconds by Hera Leto system, which is a home-based digital system
Waist circumstance | 3 months
  Using a measuring tape (cm)
Blood pressure | 3 months
  Using a sphygmomanometer (mmHg)
Concentration of high density lipoprotein cholesterol (HDL) | 3 months
  Through blood test (mg/dL)
Concentration of blood glucose | 3 months
  Through blood test (mmol/L)
Concentration of triglycerides | 3 months
  Through blood test (mg/dL)
Visceral fat area | 3 months
  Measured by bioelectrical Impedance Analysis (Tanita) in units of area (cm2)
Chinese version of the Pittsburgh sleep quality questionnaire | 3 months
  measured by 19-item scale, a range of 0-21; higher scores indicate worse sleep quality)
Chinese version of WHO self-care scale | 3 months
  6-item scale for measuring self-care capacity; a range of 6 to 18, with a higher score indicating low self-care ability
Chinese version of Geriatric Depression Scale | 3 months
  15-item scale for measuring depression; a range of 0-15; a score of >5 indicating depression
Chinese version of the Perceived Stress Scale | 3 months
  14-item scale for measuring stress level; a range from 0 to 56; a higher score indicates more perceived stress
Wong-Baker Face Pain Rating Scale | 3 months
  it measures pain severity with a range from 0 to 10
The Chinese version of the Brief Pain Inventory | 3 months
  It has 9 items measuring pain intensity
Chinese version of Medical Outcomes Study Social Support Survey | 3 months
  20-item, with a score ranging from 0 to 100, with a higher score indicating better perceived social support.
Chinese version of the General Self-efficacy Scale | 3 months
  10-item scale with a range from 10 to 40, with a higher score indicating more self-efficacy
Digital Health Literacy Scale | 3 months
  8-item scale with a range from 8 to 40, with higher scores indicating higher perceived eHealth literacy)
Chinese version of the Five facet mindfulness questionnaire | 3 months
  20-item scale; each facet score is the average of the four items, ranging from 1 to 5, with higher scores indicating higher mindfulness levels
Mindfulness | 3 months
  30-item Chinese version of Nonattachment Scale (a total mean score from 0 to 6, with a higher average score corresponding to higher nonattachment)
Chinese version of Self-compassion Scale Short-Form | 3 months
  12-item scale; a total score between 16 and 80, a higher score indicating higher self-compassion)
Chinese version of Sense of Coherence Scale | 3 months
  13-item scale; a total score range from 13 to 91,a higher score indicating a stronger sense of coherence)

CONTACTS AND LOCATIONS:
Locations (1):
- Yan Chai Hospital Social Services Department, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No